CLINICAL TRIAL: NCT04110587
Title: Hyaluronic Acid Evaluation as Adjuvant to Temporomandibular Joint Arthroscopy in Wilkes Stages
Brief Title: Hyaluronic Acid Evaluation as Adjuvant to Temporomandibular Joint Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DUROLANE2013
Record Dates: First submitted 2019-09-23; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Temporomandibular Joint Disc Displacement; Temporomandibular Joint Disorders
Keywords: hyaluronic acid; temporomandibular joint arthroscopy; internal derangements; disc displacement; temporomandibular disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Hyaluronic Acid; Anti-Infective Agents; Adrenal Cortex Hormones; Anti-Inflammatory Agents; Analgesics; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment allocation was concealed from participants and examiner (using sealed and numbered opaque envelopes by the research coordinator), and the data analyst (by encoded data).

ARMS (2):
- arthroscopy (Placebo Comparator): Temporomandibular joint arthroscopy is performed under general anesthesia by the same expert temporomandibular joint arthroscopy surgeon. Lysis and Lavage is performed in the upper joint space in all cases. Ringer's lactate is use as irrigation fluid. All participants receive Amoxicillin / Clavulanic Acid, 1g I.V. and Dexamethasone, 4 mg I.V. (Intraoperative); as well as Amoxicillin / clavulanic acid, 500/125 mg / 8h / 5 days by mouth; Diclofenac 100 mg / 12h / 5 days by mouth; and Metamizol 575 mg / 8h by mouth (Post-operatively). Soft diet and a home exercise program are implemented in all patients after 24 hours post-operative.
  Interventions: Procedure: Temporomandibular Joint Arthroscopy; Drug: Antibiotic therapy; Drug: corticosteroid; Drug: Antiinflammatories; Drug: Analgesics; Other: Exercise program
- arthroscopy plus hyaluronic Acid (Active Comparator): Temporomandibular joint arthroscopy is performed under general anesthesia by the same expert temporomandibular joint arthroscopy surgeon. Lysis and Lavage is performed in the upper joint space in all cases. Ringer's lactate is use as irrigation fluid. All participants receive Amoxicillin / Clavulanic Acid, 1g I.V. and Dexamethasone, 4 mg I.V. (Intraoperative); as well as Amoxicillin / clavulanic acid, 500/125 mg / 8h / 5 days by mouth; Diclofenac 100 mg / 12h / 5 days by mouth; and Metamizol 575 mg / 8h by mouth (Post-operatively). Soft diet and a home exercise program are implemented in all patients after 24 hours post-operative. An hyaluronic acid injection of 1 mL (Durolane®, 20 mg / mL, Zambon, Barcelona, Spain) at the end of arthroscopy that was only performed in this arm.
  Interventions: Biological: Hyaluronic Acid; Procedure: Temporomandibular Joint Arthroscopy; Drug: Antibiotic therapy; Drug: corticosteroid; Drug: Antiinflammatories; Drug: Analgesics; Other: Exercise program

INTERVENTIONS:
Biological: Hyaluronic Acid — 1 mL Hyaluronic Acid Injection (20 mg/mL, 7000 KDa) at the end of arthroscopy .
  Other Names: Sodium Hyaluronate
  Arms: arthroscopy plus hyaluronic Acid
Procedure: Temporomandibular Joint Arthroscopy — Lysis and Lavage
Drug: Antibiotic therapy — Amoxicillin / Clavulanic Acid, 1g I.V. (Intraoperative); as well as Amoxicillin / clavulanic acid, 500/125 mg / 8h / 5 days by mouth (Post-operative).
Drug: corticosteroid — Dexamethasone, 4 mg I.V. (Intraoperative)
Drug: Antiinflammatories — Diclofenac 100 mg / 12h / 5 days by mouth (Post-operatively).
Drug: Analgesics — Metamizol 575 mg / 8h by mouth (Post-operatively)
Other: Exercise program — Home exercise program

SUMMARY:
This study evaluates the addition of hyaluronic acid to temporomandibular joint arthroscopy in the treatment of internal derangements in adults. A participants group will receive temporomandibular joint arthroscopy plus hyaluronic acid, while the other group will receive temporomandibular joint arthroscopy. Hypothesis: hyaluronic acid as an adjunct in temporomandibular joint arthroscopic surgery provides additional benefits in clinical and radiological outcomes in temporomandibular joint internal derangements.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of temporomandibular joint internal derangements in Wilkes stages III and IV by magnetic resonance imaging
* Limitation of maximum oral opening or duplication of joint pain by palpation
* lack of response to conservative therapies

Exclusion Criteria:

* Any degenerative systemic disease of muscular or joint involvement (rheumatoid arthritis, etc.)
* Previous temporomandibular joint surgical treatment: arthrocentesis, arthroscopy or open surgery
* Infection in Temporomandibular Joint or in puncture site
* Hyaluronic acid or corticosteroids injection in Temporomandibular Joint in previous 6 months
* Pregnant or breastfeeding women
* Participants who refuse to complete the treatment or unavailable to complete the follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-12-10 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Pain Scores on the Visual Analog Scale at 3,6,9 and 12 Months | From enrollment to end of study at 12 Months. Baseline, Month 3, Month 6, Month 9, Month 12.
  Visual Analog Scale 0 to 10. Higher values represent a worse outcome.
Mean Change from Baseline in Maximal Oral Opening Scores (mm) at 3,6,9 and 12 Months | From enrollment to end of study at 12 Months. Baseline, Month 3, Month 6, Month 9, Month 12.
  measured from edge of upper central incisor to edge of lower antagonist incisor. Range scale 0 to 60 (mm). Higher values represent a better outcome.
Mean Change from Baseline in Oral Health Impact Profile-14 Spanish Version (OHIP-14sp) questionnaire Scores at 6 and 12 Months | From enrollment to end of study at 12 Months. Baseline, Month 6, Month 12.
  OHIP-14sp questionnaire total average score to measure Oral Health-Related Quality of Life. Range scale 0 to 56. Higher values represent a worse outcome. Total average score is calculated by adding the score of each question and dividing by 14

SECONDARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events | From intervention to end of study at 12 Months. During procedure or immediately after intervention, Month 3, Month 6, Month 9, Month 12.
  any adverse response to the intervention
Symptoms Duration Mean (Months) | At baseline
  symptoms duration mean reported by the participants
Number of Participants with chondromalacia | During intervention
  arthroscopic finding
Number of Participants with synovitis | During intervention
  arthroscopic finding
Irrigation Volume Mean (cc) | During intervention
  average irrigation fluid used during intervention
Number of Participants with Occlusal Stabilization Splint | From enrollment to end of study at 12 Months. Baseline, Month 3, Month 6, Month 9, Month 12.
  stabilization splint use reported by the participant
Number of Participants with Osteophyte by magnetic resonance imaging | At baseline and Month 12.
  radiographic finding in jaw condyle
Number of Participants with joint surfaces flattening by magnetic resonance imaging | At baseline and Month 12
  radiographic finding in jaw condyle or temporal bone
Number of Participants with Subchondral Geode by magnetic resonance imaging | At baseline and Month 12
  radiographic finding in jaw condyle
Disc Position by magnetic resonance imaging | At baseline and Month 12
  No Displacement, Disc Displacement with Reduction, Disc Displacement without Reduction
Number of Participants with pain in masseter muscle by digital palpation | From enrollment to end of study at 12 Months. Baseline, Month 3, Month 6, Month 9, Month 12.
  pain reported by the participant
Number of Participants with pain in Temporal muscle by digital palpation | From enrollment to end of study at 12 Months. Baseline, Month 3, Month 6, Month 9, Month 12.
  pain reported by the participant
Number of Participants with pain in Medial Pterygoid Muscle by digital palpation | From enrollment to end of study at 12 Months. Baseline, Month 3, Month 6, Month 9, Month 12.
  pain reported by the participant
Number of Participants with pain in digastric Muscle by digital palpation | From enrollment to end of study at 12 Months. Baseline, Month 3, Month 6, Month 9, Month 12.
  pain reported by the participant
Number of Participants with pain in Genihyoid Muscle by digital palpation | From enrollment to end of study at 12 Months. Baseline, Month 3, Month 6, Month 9, Month 12.
  pain reported by the participant
Number of Participants with pain in Mylohyoid Muscle by digital palpation | From enrollment to end of study at 12 Months. Baseline, Month 3, Month 6, Month 9, Month 12.
  pain reported by the participant

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cano Sánchez, Study Director — Universidad Complutense de Madrid; Julian Campo Trapero, Study Director — Universidad Complutense de Madrid; Mario Fernando Muñoz Guerra, Study Director — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Oscar Gabriel Castaño Joaqui, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montero-Martin J, Bravo-Perez M, Albaladejo-Martinez A, Hernandez-Martin LA, Rosel-Gallardo EM. Validation the Oral Health Impact Profile (OHIP-14sp) for adults in Spain. Med Oral Patol Oral Cir Bucal. 2009 Jan 1;14(1):E44-50. PMID 19114956
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981
- [Background] Shi Z, Guo C, Awad M. Hyaluronate for temporomandibular joint disorders. Cochrane Database Syst Rev. 2003;(1):CD002970. doi: 10.1002/14651858.CD002970. PMID 12535445
- [Background] Wilkes CH. Internal derangements of the temporomandibular joint. Pathological variations. Arch Otolaryngol Head Neck Surg. 1989 Apr;115(4):469-77. doi: 10.1001/archotol.1989.01860280067019. PMID 2923691
- [Derived] Castano-Joaqui OG, Cano-Sanchez J, Campo-Trapero J, Munoz-Guerra MF. TMJ arthroscopy with hyaluronic acid: A 12-month randomized clinical trial. Oral Dis. 2021 Mar;27(2):301-311. doi: 10.1111/odi.13524. Epub 2020 Jul 25. PMID 32609918